CLINICAL TRIAL: NCT00821327
Title: Phase II Trial of Gemcitabine, Cisplatin, and Sunitinib in Patients With Advanced/Metastatic Urothelial Carcinoma
Brief Title: Gemzar, Cisp, Sunitinib Urothelial Ca
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06040; WS356467 (Other: Pfizer)
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — Gemcitabine; Cisplatin; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Arm (Experimental): Gemcitabine, Cisplatin, Sunitinib
  Interventions: Drug: Gemcitabine, Cisplatin, Sunitinib

INTERVENTIONS:
Drug: Gemcitabine, Cisplatin, Sunitinib — Patients will receive gemcitabine 800 mg/m2 IV (Days 1 and 8), cisplatin 60 mg/m2 IV (Day 1), and sunitinib 37.5 mg PO daily (Days 1-14) of each 21-day cycle.
  2. One cycle of treatment is defined as 21 days (3 weeks). Restaging studies will be performed after every 3 cycles of therapy.
  3. Successive cycles will be initiated every 3 weeks, and will be continued through 6 cycles unless a patient shows evidence of disease progression or intolerable toxicity.
  Other Names: Gemzar, Sutent

SUMMARY:
The primary objective of this nonrandomized Phase II study is to evaluate the objective response rate (ORR, CR+PR) in patients with advanced/metastatic UC treated with the combination of gemcitabine, cisplatin, and sunitinib.

DETAILED DESCRIPTION:
Given the strong preclinical rationale for targeting angiogenesis in urothelial carcinoma (UC), the evidence supporting co-targeting of VEGFR2 and PDGF, the safety and efficacy of single-agent sunitinib in patients with UC, and preclinical evidence of synergy with the combination of sunitinib and cisplatin, the evaluation of sunitinib in combination with gemcitabine plus cisplatin in previously untreated patients with metastatic UC is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Has histological documentation of diagnosis of transitional cell carcinoma (TCC) of the bladder, urethra, ureter, or renal pelvis (histology may be mixed, but still requires a component of TCC; measurable disease only)
2. Has unresectable or metastatic disease
3. Has a Karnofsky Performance Status greater than or equal 60 percent
4. Is 18 years of age or older
5. Has laboratory values as defined by the protocol
6. Has resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to NCI CTCAE (v3.0) Grade less than or equal to 1
7. Has normal cardiac function as evidenced by a LVEF greater than or equal to 50 percent, as determined by multiple gated acquisition (MUGA) scan or an echocardiogram (ECHO). The same method must be used throughout the study to evaluate LVEF.
8. Has a negative serum pregnancy test within 7 calendar days prior to registration (female patients of childbearing potential [not surgically sterilized and between menarche and 1 year postmenopausal])
9. Is not currently breastfeeding
10. If fertile, patient (male or female) has agreed to use an acceptable method of birth control to avoid pregnancy for the duration of the study and for a period of 3 months thereafter.
11. Has signed a Patient Informed Consent Form, Has signed a Patient Authorization Form

Exclusion Criteria:

1. Has had prior treatment with systemic chemotherapy (prior intravesical therapy is permitted)
2. Has had major surgery or radiation therapy within 4 weeks of starting the study treatment
3. Has had NCI CTCAE (Version 3.0) Grade 3-4 hemorrhage within 4 weeks of starting the study treatment
4. Has a history of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan. However treated, stable and asymptomatic brain metastases are allowed.
5. Has had any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
6. Has ongoing cardiac dysrhythmias of NCI CTCAE (Version 3.0) Grade 2
7. Has prolonged QTc interval on baseline EKG
8. Has uncontrolled hypertension (grater than 150/100 mm Hg despite optimal medical therapy)
9. Has pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
10. Has known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
11. Is receiving concomitant use of any other investigational drugs or has received such drug within 28 days prior to registration
12. Is receiving concurrent treatment on another clinical trial, including supportive care
13. Has ongoing treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg PO daily for thromboembolic prophylaxis allowed). Patients on warfarin (greater than 2mg) for thrombosis must be switched to low molecular weight heparin (ie, Lovenox), prior to registration for protocol therapy.
14. Is currently taking drugs having proarrhythmic potential (terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide and flecainide) within 7 days prior to Day 1 of Cycle 1 (dosing) (and throughout study)
15. Is currently on CYP3A4 inhibitors (see Section 5) within 7 days prior to Day 1 of Cycle 1 (dosing), with the exception of amiodarone, which should be discontinued within 6 months prior to Day 1 of Cycle 1 (dosing)
16. Is currently on CYP3A4 inducers (see Section 5) within 14 days prior to Day 1 of Cycle 1 (dosing)
17. Has been taking herbal or alternative medications within the past 7 days or refuses to discontinue the use of herbal or alternative therapies within 7 days prior to Day 1 of Cycle 1 (dosing)
18. Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection
19. Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix), which could affect the diagnosis or assessment of any of the study drugs.
20. Is a pregnant or nursing woman. Patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the Study Investigator or Treating Physician. Male patients must be surgically sterile or agree to use effective contraception.

Is unable to comply with requirements of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guru Sonpavde, MD, Principal Investigator — US Oncology; Thomas E Hutson, DO, Principal Investigator — US Oncology
Locations (48):
- United States (48):
  - Arizona Oncology Associates, Tucson, Arizona
  - Advanced Medical Specialties, Miami, Florida
  - Florida Cancer Institute - New Hope, New Port Richey, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Alliance Hematology Oncology PA., Westminster, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Arch Medical Services, Inc., Saint Louiis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hematology-Oncology Associates of Northern NJ, PA, Morristown, New Jersey
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Willamette Valley Cancer Center, Springfield, Oregon
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Cancer Center - Abilene, Abilene, Texas
  - Texas Oncology, P.A. -Amarillo, Amarillo, Texas
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology - Round Rock Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Texas Oncology, Beaumont, Texas
  - Texas Oncology, P.A. - Bedford, Bedford, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology/Methodist Charlton Cancer Ctr., Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Center - East, El Paso, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology, Garland, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center, McAllen, Texas
  - Texas Oncology, PA, Allison Cancer Center, Midland, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Cancer Care Centers of South Texas-HOAST, San Antonio, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology Cancer Center - Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Salem, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Pudget Sound Cancer Center, Edmonds, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington

REFERENCES:
- [Derived] Galsky MD, Hahn NM, Powles T, Hellerstedt BA, Lerner SP, Gardner TA, Yu M, O'Rourke M, Vogelzang NJ, Kocs D, McKenney SA, Melnyk AM Jr, Hutson TE, Rauch M, Wang Y, Asmar L, Sonpavde G. Gemcitabine, Cisplatin, and sunitinib for metastatic urothelial carcinoma and as preoperative therapy for muscle-invasive bladder cancer. Clin Genitourin Cancer. 2013 Jun;11(2):175-81. doi: 10.1016/j.clgc.2012.10.001. Epub 2012 Dec 8. PMID 23228446

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm: Advanced/Metastatic UC: Gemcitabine, Cisplatin, Sunitinib
  Gemcitabine, Cisplatin, Sunitinib: Patients will receive gemcitabine 800 mg/m2 IV (Days 1 and 8), cisplatin 60 mg/m2 IV (Day 1), and sunitinib 37.5 mg PO daily (Days 1-14) of each 21-day cycle.
  2. One cycle of treatment is defined as 21 days (3 weeks). Restaging studies will be performed after every 3 cycles of therapy.
  3. Successive cycles will be initiated every 3 weeks, and will be continued through 6 cycles unless a patient shows evidence of disease progression or intolerable toxicity.
Period: Overall Study
Arm/Group | Study Arm: Advanced/Metastatic UC
Started | 36
Completed | 1
Not Completed | 35
Not completed — Adverse Event | 13
Not completed — Patient Request | 1
Not completed — Investigator Request | 2
Not completed — Sponsor Request | 1
Not completed — Disease Progression | 13
Not completed — Other/Unknown | 5

BASELINE CHARACTERISTICS:
Arm/Group | Study Arm: Advanced/Metastatic UC
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 32
  Hispanic | 2
  Asian | 1
  Black | 1
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR, CR+PR) in Patients With Advanced/Metastatic UC Treated With the Combination of Gemcitabine, Cisplatin, and Sunitinib.
Description: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: 2 years
Population: All eligible patients who meet the protocol-specified efficacy analyses requirements and who have received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Study Arm: Advanced/Metastatic UC
Number analyzed (Participants) | 33
Percentage of participants | 48.5 [30.8 to 66.5]

2. Secondary Outcome: Progression-free Survival
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
  Progression (PD) is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: 2 years
Population: ITT population
Measure: Median (Full Range); unit: Month
Arm/Group | Study Arm: Advanced/Metastatic UC
Number analyzed (Participants) | 36
Month | 8.0 [7.0 to 14.0]

3. Secondary Outcome: Ovarall Survival (OS)
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 2 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Study Arm: Advanced/Metastatic UC
Number analyzed (Participants) | 36
months | 13.8 [10.1 to 22.9]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | Study Arm: Advanced/Metastatic UC
Serious Adverse Events (participants affected / at risk) | 7/33
Other Adverse Events (participants affected / at risk) | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm: Advanced/Metastatic UC (N=33)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
BLOOD PRESSURE INCREASED (Blood and lymphatic system disorders) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
HEMOGLOBIN DECREASED (Blood and lymphatic system disorders) | 1 (1)
LYMPHADENOPATHY THORACIC (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
PANCREATITIS (Infections and infestations) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm: Advanced/Metastatic UC (N=33)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3)
ALT INCREASED (Metabolism and nutrition disorders) | 2 (5)
ANEMIA (Blood and lymphatic system disorders) | 22 (78)
ANOREXIA (Gastrointestinal disorders) | 8 (8)
AST INCREASED (Metabolism and nutrition disorders) | 2 (6)
BLEEDING NOSE (Blood and lymphatic system disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 9 (10)
CREATININE CLEARANCE DECREASED (Metabolism and nutrition disorders) | 2 (2)
CREATININE SERUM INCREASED (Metabolism and nutrition disorders) | 3 (4)
DEHYDRATION (Gastrointestinal disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 6 (10)
DIZZINESS (Nervous system disorders) | 2 (3)
EDEMA (Blood and lymphatic system disorders) | 2 (2)
FATIGUE (General disorders) | 18 (34)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 9 (9)
HAND-FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 3 (3)
HEADACHE (Nervous system disorders) | 2 (2)
HEMATURIA (Renal and urinary disorders) | 2 (2)
HICCUP (Gastrointestinal disorders) | 2 (2)
HYPERTENSION (Cardiac disorders) | 5 (8)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 3 (5)
INSOMNIA (General disorders) | 3 (4)
LEUCOPENIA (Blood and lymphatic system disorders) | 10 (40)
MUCOSAL SORES (Infections and infestations) | 2 (2)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 16 (22)
NEUROPATHY (Nervous system disorders) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 30 (113)
PAIN (General disorders) | 4 (5)
RASH (Skin and subcutaneous tissue disorders) | 4 (6)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 7 (8)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 24 (88)
VOMITING (Gastrointestinal disorders) | 7 (9)
WEIGHT LOSS (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No